CLINICAL TRIAL: NCT04877561
Title: Translation, Trans-cultural Adaptations and Test-retest Reliability of the Headache Disability Questionnaire (HDQ)
Brief Title: Test-Retest Reliability of the German Version of the Headache Disability Questionnaire (HDQ).
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Zurich University of Applied Sciences (Other)
Responsible Party: Principal Investigator, Markus J. Ernst, Research fellow, MSc,, Zurich University of Applied Sciences
Other Study IDs: ZUAS HDQ
Record Dates: First submitted 2021-05-03; First posted 2021-05-07 (Actual); Last update posted 2021-05-12 (Actual); Status verified 2021-05

CONDITIONS: Headache Disorders
MeSH Terms: conditions — Headache Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
a translated and cultural adapted version of the HDQ will be tested on two occasions with headache patients who are currently in physiotherapeutic treatment due to their headache condition

DETAILED DESCRIPTION:
The test-retest reliability of the German version of the HDQ will be tested to assess the reproducibility of the test results with a stable condition of the participants over a short period of time. For this purpose, it is planned to administer the questionnaire twice in row at an interval of 48 - 72 hours to headache patients in outpatient physiotherapy. The chosen setting limits the sample to a common intervention measure (physiotherapy), so that primary and secondary headache types can be included and the requirements of the original study can be maintained. In the period between the two tests, subjects should not receive physiotherapy, because it can often have different effects on headache. This can lead to uneven changes in the sample and affect the variance of the test results. However, subjects are allowed to take their usual medications. To avoid recall bias, an online survey tool (RedCAP) to conduct the questionnaire will be used. It is designed so that, only one question appears per slide, no overview of responses is allowed and the questions are displayed in a different order at the second testing. The lower prevalence of headaches after the age of 65 years is taken into account in the inclusion criteria.

ELIGIBILITY:
Inclusion Criteria:

* within physiotherapeutic care due to headache for no longer than 3 months
* headache conditions for at least one month and at least once /month
* live in Switzerland
* give informed consent

Exclusion Criteria:

* not in physiotherapeutic care
* in physiotherapeutic care due to other conditions not associated with headache
* younger than 18 and older than 65 years

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects suffering from a headache condition and are due to that in physiotherapeutic care
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2021-06-01 (Estimated); Primary Completion 2022-07-31 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
Headache | June 21 to July 22
  Nine item headache disability questionnaire (HDQ)

SECONDARY OUTCOMES:
Headache disorder | June 21 to July 22
  Migraine, Tension-type headache, other

CONTACTS AND LOCATIONS:
Overall Officials: Markus J Ernst, Master, Study Director — Zurich University of Applied Sciences
Locations (1):
- Zurich University of Applied Sciences, Winterthur, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No
There is no intention to share the IPD

REFERENCES:
- [Background] Niere K, Quin A. Development of a headache-specific disability questionnaire for patients attending physiotherapy. Man Ther. 2009 Feb;14(1):45-51. doi: 10.1016/j.math.2007.09.006. Epub 2007 Nov 7. PMID 17997346
- [Background] Stovner LJ, Andree C. Prevalence of headache in Europe: a review for the Eurolight project. J Headache Pain. 2010 Aug;11(4):289-99. doi: 10.1007/s10194-010-0217-0. Epub 2010 May 16. PMID 20473702
- [Background] Luedtke K, Basener A, Bedei S, Castien R, Chaibi A, Falla D, Fernandez-de-Las-Penas C, Gustafsson M, Hall T, Jull G, Kropp P, Madsen BK, Schaefer B, Seng E, Steen C, Tuchin P, von Piekartz H, Wollesen B. Outcome measures for assessing the effectiveness of non-pharmacological interventions in frequent episodic or chronic migraine: a Delphi study. BMJ Open. 2020 Feb 12;10(2):e029855. doi: 10.1136/bmjopen-2019-029855. PMID 32051295
- [Background] Benz T, Lehmann S, Gantenbein AR, Sandor PS, Stewart WF, Elfering A, Aeschlimann AG, Angst F. Translation, cross-cultural adaptation and reliability of the German version of the migraine disability assessment (MIDAS) questionnaire. Health Qual Life Outcomes. 2018 Mar 9;16(1):42. doi: 10.1186/s12955-018-0871-5. PMID 29523138
- [Background] Marx RG, Menezes A, Horovitz L, Jones EC, Warren RF. A comparison of two time intervals for test-retest reliability of health status instruments. J Clin Epidemiol. 2003 Aug;56(8):730-5. doi: 10.1016/s0895-4356(03)00084-2. PMID 12954464